CLINICAL TRIAL: NCT04887870
Title: A Multicenter, Open-label Rollover Study of Sitravatinib Alone or in Combination With Other Anticancer Therapies in Patients With Advanced or Metastatic Solid Malignancies
Brief Title: Study of Sitravatinib With or Without Other Anticancer Therapies Receiving Clinical Benefit From Parent Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA248-0003; CA248-0003 (Other: Bristol-Myers Squibb Protocol ID); 516-014 (Other: Mirati Therapeutics Protocol ID)
Record Dates: First submitted 2021-04-28; First posted 2021-05-14 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Advanced or Metastatic Solid Malignancies
MeSH Terms: interventions — sitravatinib; Nivolumab; pembrolizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 2/3: Open label extension of parent study (Experimental): The current study is designed to allow continued access to sitravatinib and to evaluate the safety and tolerability of sitravatinib alone or in combination with other anticancer therapies in patients who are deriving clinical benefit in a previous parent clinical trial.
  Interventions: Drug: Sitravatinib; Drug: Nivolumab; Drug: Pembrolizumab; Drug: Enfortumab Vedotin-Ejfv; Drug: Ipilimumab

INTERVENTIONS:
Drug: Sitravatinib — Sitravatinib is a small molecule inhibitor of receptor tyrosine kinases.
  Other Names: MGCD516
Drug: Nivolumab — Nivolumab is a programmed death receptor-1 (PD-1) blocking antibody
  Other Names: OPDIVO
Drug: Pembrolizumab — Pembrolizumab is a programmed death receptor-1 (PD-1) blocking antibody
  Other Names: KEYTRUDA
Drug: Enfortumab Vedotin-Ejfv — Enfortumab is a Nectin-4 directed antibody-drug conjugate (ADC) comprised of a monoclonal antibody conjugated to the small molecule microtubule disrupting agent, monomethyl auristatin E (MMAE)
  Other Names: PADCEV
Drug: Ipilimumab — Ipilimumab is a CTLA-4 (cytotoxic T-lymphocyte-associated protein 4) blocking antibody
  Other Names: YERVOY

SUMMARY:
A Study of Sitravatinib Alone or in Combination with Other Anticancer Therapies in Advanced or Metastatic Malignancies

DETAILED DESCRIPTION:
Sitravatinib is a spectrum-selective receptor tyrosine kinase (RTK) inhibitor that inhibits several closely related RTKs including the TAM family (Tyro3/Axl/MERTK), VEGFR2, KIT, and MET.

The current study is designed to allow continued access to sitravatinib and to evaluate the safety and tolerability of sitravatinib alone or in combination with other anticancer therapies in patients who are deriving clinical benefit in a previous parent clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Currently receiving sitravatinib single- agent or in combination with other therapeutic agent(s) in another Mirati- sponsored protocol
* Currently tolerating the treatment regimen in the parent protocol
* Experiencing clinical benefit with or without prior radiographic progression from the treatment regimen in the parent protocol in the opinion of the investigator and the investigator determines that continuing treatment is in the patient's best interest

Exclusion Criteria:

* Known or suspected presence of other cancer
* Other life- threatening illness or organ system dysfunction compromising safety evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-09-25 (Actual)

PRIMARY OUTCOMES:
Frequency of subjects experiencing treatment-related AEs. | 24 Months
  Frequency of subjects experiencing treatment-related AEs.

SECONDARY OUTCOMES:
Time to clinical or radiographic progression on study. | 24 Months
  Time to clinical or radiographic progression on study.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- United States (13):
  - Rocky Mountain Cancer Centers - Littleton, Littleton, Colorado
  - Local Institution - 516-014-029, Goshen, Indiana
  - Local Institution - 516-014-002, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Local Institution - 516-014-005, Minneapolis, Minnesota
  - Urology Cancer Center and GU Research Network, Omaha, Nebraska
  - Local Institution - 516-014-011, Albany, New York
  - Memorial Sloan Kettering Cancer Center - Arnold and Marie Schwartz Cancer Research Building, New York, New York
  - Local Institution - 516-014-004, Columbus, Ohio
  - Local Institution - 516-014-001, Austin, Texas
  - USOR - Texas Oncology Northeast Texas - Denison, Denison, Texas
  - Local Institution - 516-014-013, Houston, Texas
  - NEXT Virginia, Fairfax, Virginia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com